CLINICAL TRIAL: NCT01448499
Title: Clozapine Versus Amisulpride Versus Their Combination in the Treatment of Drug-resistant Schizophrenia Patients
Brief Title: Clozapine Versus Amisulpride in Treatment-resistant Schizophrenia Patients
Acronym: ClozAmi
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Geha Mental Health Center (Other)
Responsible Party: Principal Investigator, Amir Krivoy, Senior psychiatrist, Geha Mental Health Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GMCH-014-11
Record Dates: First submitted 2011-10-02; First posted 2011-10-07 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Schizophrenia; Treatment Resistant Disorders
Keywords: schizophrenia; clozapine; amisulpride; combination; treatment resistant
MeSH Terms: conditions — Schizophrenia | interventions — Clozapine; Amisulpride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Clozapine (Experimental): Clozapine monotherapy
  Interventions: Drug: Clozapine
- Amisulpride (Experimental): Amisulpride monotherapy
  Interventions: Drug: Amisulpride
- Augmentation (Experimental): Augmentation of clozapine with amisulpride
  Interventions: Drug: Clozapine+Amisulpride

INTERVENTIONS:
Drug: Clozapine — escalating dose of clozapine up to 900 mg/day
  Arms: Clozapine
Drug: Amisulpride — escalating dose of amisulpride up to 800 mg/day
  Arms: Amisulpride
Drug: Clozapine+Amisulpride — augmentation of clozapine with amisulpride
  Arms: Augmentation

SUMMARY:
Background: schizophrenia is a debilitating mental disorder affecting about 1% of the general population. About 30% of patients will not react to current drug treatment and defined as treatment-resistant schizophrenia patients (TRSP). The best studied therapeutic option for this population is clozapine therapy. Clozapine was shown to be effective than any other antipsychotic drug in TRSP. Moreover, augmentation of clozapine was not demonstrated to be more effective than clozapine monotherapy. Albeit Clozapine superiority in TRSP, its use may be involved with many adverse effects, some of them are life-threatening, and need for routine blood tests. Amisulpride is an atypical antipsychotic drug with a different mechanism of action than clozapine, with less adverse effects. No study compared directly amisulpride and clozapine in TRSP.

Study objective: to compare, for the first time, the broad clinical effectiveness of clozapine and amisulpride and their combination in TRSP.

Study Design: a clinical, prospective, naturalistic, randomized, comparative study simulating a real-world approach of clinical decision making.

Methods: a total of 140 TRSP will be recruited from a large regional mental health center. Participants will be randomized into two treatment groups (70 in each group): clozapine monotherapy and amisulpride monotherapy. Assessment will be done following 10 and 20 weeks of treatment. In case of treatment failure (insufficient clinical response or severe adverse effect) participants will be offered either to switch to clozapine treatment (for failed amisulpride treatment) or to augment clozapine with amisulpride (for failed clozapine monotherapy patients). Thereafter, participants will be followed-up for a year. Assessment will be made using clinician rated scales and self-completed questionnaires, rating the broad phenomenology of schizophrenia (psychosis, mood, anxiety, obsessive-compulsive, cognitive and quality of life) and drug-related adverse effects (objective and subjective).

Analysis: comparison of the effectiveness of the three treatment groups: amisulpride, clozapine and their combination, in the various dimensions of TRSP.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of schizophrenia according to DSM-IV-TR criteria
2. Treatment-resistant schizophrenia, defined as: documented treatment failure (insufficient clinical response or severe adverse effects) of two antipsychotics (one of them should be atypical) for an adequate duration of 6 weeks and in a sufficient dose of at least 600 mg/day of chlorpromazine equivalent
3. Age 18-65 years
4. Basal PANSS > 75
5. CGI-S >3
6. Persistent positive psychotic symptoms, with rating scores of moderate or worse on at least two of four positive symptom items (delusions, conceptual disorganization, hallucinatory behavior, and suspiciousness/persecution) on Positive and Negative Syndrome Scale (PANSS).
7. Competent and willing to provide written, informed consent

Exclusion Criteria:

1. Patients with concomitant treatment with lithium, anticonvulsants, antidepressants
2. Patients with underlying severe medical illness, such as cardiovascular disease, cerebrovascular disease, bone marrow suppression or epilepsy
3. A previous trial of clozapine or amisulpride
4. Any known contraindication for treatment with clozapine or amisulpride
5. Any woman who is pregnant or planning a pregnancy, and any woman of child bearing potential unless using adequate contraception

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-10; Primary Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Positive and Negative Syndrome Scale (PANSS) | 10, 20 weeks and endpoint

SECONDARY OUTCOMES:
Change from baseline in Clinical Global Impression - Severity (CGI-S) | 10 , 20 weeks and endpoint
Change from baseline in Beck Depression Inventory (BDI) | 10 , 20 weeks and endpoint
Change from baseline in Beck Anxiety Inventory (BAI) | 10, 20 weeks and endpoint
Change from baseline in Schizophrenia Quality of Life Scale (SQLS) | 10, 20 weeks and endpoint
Change from baseline in Simpson-Angus Scale (SAS) | 5, 10, 15, 20 weeks, endpoint
Change from baseline in Clozapine Adverse Effects Inventory (CAEI) | 5, 10 ,15, 20 weeks, endpoint

CONTACTS AND LOCATIONS:
Locations (1):
- Geha Mental Health Center, Petah Tikva, Israel